CLINICAL TRIAL: NCT03947736
Title: Detection of HER2 Amplification Status and Dynamic Monitoring of Specific Mutations in Patients With Recurrent or Metastatic Breast Cancer by Digital PCR
Brief Title: Dynamic Monitoring of HER2 and ctDNA Specific Mutations in Patients With Recurrent or Metastatic Breast Cancer by Digital PCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Questgenomics (Other)
Responsible Party: Principal Investigator, Peng Yuan, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: NCC1824
Record Dates: First submitted 2019-05-10; First posted 2019-05-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Recurrent or Metastatic Breast Cancer
MeSH Terms: conditions — Recurrence; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with positive HER2 amplification
  Interventions: Diagnostic Test: cfDNA was detected by dPCR
- patients with negative HER2 amplification
  Interventions: Diagnostic Test: cfDNA was detected by dPCR

INTERVENTIONS:
Diagnostic Test: cfDNA was detected by dPCR — Without drug intervention, the patient's peripheral blood was collected and cfDNA was extracted for digital PCR detection.

SUMMARY:
This was a prospective, single-center clinical study. The study was designed to investigate the relationship between plasma HER2 amplification or specific mutations abundance and clinical response in patients with recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
Patients were divided into two groups according to ctDNA HER2 amplification status by dPCR method. Group A consisted of patients with positive HER2 amplification at the time of enrollment. Plasma HER2 amplification status was measured by dPCR during dynamic monitoring. GroupB consists of patients with negative HER2 amplification when enrolled. Plasma samples were collected before treatment and breast cancer hotspot mutations were detected with NGS, According to the NGS test results, patient's specific mutations were analyzed and selected, which and plasma HER2 amplification status were measured by dPCR during dynamic monitoring.

The study was designed to investigate the relationship between plasma HER2 amplification or specific mutations abundance and imaging assessment in patients with recurrent or metastatic breast cancer. And also to investigate the proportion of predicting in advance the treatment efficacy of recurrent or metastatic breast cancer by plasma HER2 ctDNA, as well as the median time difference between predicted clinical efficacy by changes in abundance of plasma HER2 amplification specific mutations and medical imaging evaluation in patients.

The study only focus on ctDNA detection and does not involve any interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed by pathology and/or histology/cytology as breast cancer;
2. Patients with recurrent or metastatic breast cancer who are 18 to 75 years old, not limited to the first relapse or metastasis;
3. There are evaluable tumor lesions;
4. Physical strength: ECOG score 0-1;
5. The expected survival period is more than 3 months;
6. Agree to be collected tissue specimen;
7. The patient has no major organ dysfunction, agrees and can implement a treatment plan based on the patient's condition.
8. Voluntary enrollment, good compliance, can be followed up and observed.

Exclusion Criteria:

1. Severe vital organs (heart, liver, kidney) dysfunction; clinically significant heart disease, classified by New York Heart Association (NYHA) as grade III-IV heart failure or more severe congestive heart failure or severe Arrhythmia requiring drug intervention; uncontrolled angina, uncontrolled arrhythmia or uncontrollable hypertension, electrocardiogram (ECG)-confirmed myocardial infarction within 6 months;
2. Have a history of organ transplantation, splenectomy;
3. Patients with other malignancies, except cured non-melanoma skin cancer, cervical carcinoma in situ, or other tumors that have been cured for at least 5 years;
4. Moderate or severe renal impairment [creatinine clearance equal to or lower than 50ml/min (calculated according to Cockroft and Gault equations)], or serum creatinine > normal upper limit (ULN); pulmonary function test FEV1 < 50% of estimated value;
5. Parallel surgical treatment of other diseases is required;
6. Patients who are pregnant or breast-feeding (women of childbearing age need to be examined for pregnancy); women of childbearing age must take contraceptive measures that the investigator considers effective;
7. Patients with or showing signs of disseminated spongiform encephalopathy or family members have the disease;
8. In the active period of other acute infectious diseases or chronic infectious diseases;
9. Have uncontrolled epilepsy, central nervous system disease or a history of mental disorders;
10. People with disabilities or with no legal capacity or legal capacity is limited;
11. Those who received a research medication or formulation/treatment (ie, participated in other trials) within 4 weeks prior to enrollment;
12. Other situations when the investigators believe that patients should not participate in this trial.

Quitting criteria:

1. The patient suffers from other diseases and needs to be immediately taken to other therapists, and is no longer suitable for sampling test;
2. Diagnosis of encephalitis and other inflammatory neuropathies;
3. After the enrollment, it is clearly determined that the subject does not meet the requirements of the subject;
4. The investigator believes that the withdrawal of the trial is in the best interest of the subject;
5. Pregnancy;
6. Poor compliance, two consecutive failures to accept testing as planned;
7. The patient him/herself or the researcher believes that it is medically required to be withdrawn from the study.
8. For subjects who discontinued the study early, the reason for the early withdrawal should be recorded, and the time of the last visit should be recorded, and the inspection items at the time of early termination of the study should be completed in the last visit as much as possible.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with recurrent or metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The study was designed to investigate the relationship between plasma HER2 amplification or specific mutations abundance and imaging assessment in patients with recurrent or metastatic breast cancer. | 2020-12-31
The study was designed to investigate the proportion of predicting in advance the treatment efficacy of recurrent or metastatic breast cancer by plasma HER2 ctDNA. | 2020-12-31

CONTACTS AND LOCATIONS:
Overall Officials: Dr. yuan, Prof, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided